CLINICAL TRIAL: NCT02540746
Title: Transdiagnostic Treatment for Early Stage Mental Health Problems in Youth: A Pilot Randomized Trial
Brief Title: Transdiagnostic Treatment for Early Stage Mental Health Problems in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Principal Investigator, Robert B Zipursky, MD, Psychiatrist, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-312
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Mental Disorders
Keywords: Emotional Dysregulation; Early Intervention; Youth Mental Health; Staging; Motivational Enhancement; Family Connections; Family Skills Training
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ERG Skills Training (Experimental): ERG Skills Training for 12 weeks
  Interventions: Behavioral: ERG Skills Training
- ERG Skills Training + ME (Experimental): ERG Skills Training for 12 weeks preceded by Motivational Enhancement for 4 weeks
  Interventions: Behavioral: ERG Skills Training; Behavioral: Motivational Enhancement
- ERG Skills Training + FAM (Experimental): ERG Skills Training with concurrent 12-week Family Skills Training
  Interventions: Behavioral: ERG Skills Training; Behavioral: Family Skills Training
- ERG Skills Training + ME + FAM (Experimental): ERG Skills Training with concurrent 12-week Family Skills Training preceded by Motivational Enhancement for 4 weeks
  Interventions: Behavioral: ERG Skills Training; Behavioral: Motivational Enhancement; Behavioral: Family Skills Training

INTERVENTIONS:
Behavioral: ERG Skills Training — Group-based Dialectical Behavior Therapy Skills Training for 12 weeks
Behavioral: Motivational Enhancement — Three week Motivational Enhancement group
  Arms: ERG Skills Training + ME; ERG Skills Training + ME + FAM
Behavioral: Family Skills Training — 12-week group-based family skills training using Family Connections model
  Other Names: Family Connections
  Arms: ERG Skills Training + FAM; ERG Skills Training + ME + FAM

SUMMARY:
The aim of this pilot study is to examine a brief manualized treatment, Emotional Regulation Group Skills Training (ERG ST), which has shown promise with high-risk youth presenting with a range of mental health concerns. The investigators will examine the effectiveness of a ERG ST group, as well as two additional components to which clients will be randomized: a motivational enhancement (ME) pre-treatment, and family skills treatment (FAM). This project will be the first to combine and test these modules as a transdiagnostic early intervention for youth in the early stages on mental illness. This pilot trial will answer the following questions: 1) What is the response rate to ERG ST compared to ERG ST plus FAM, and who benefits? 2) What is the response rate to a ME pre-treatment, and who benefits? 3) What is the acceptability of this treatment?

The ME pre-treatment will consist of four weekly one and a half hour sessions. The 12-week ERG ST will consist of 12 weekly two-hour sessions with 4-12 youths per group. The 12-week FAM will consist of 12 weekly two-hour sessions, with 16-20 caregivers per group. This study will use a two-stage randomization design to allow for balanced groups if there is differential attrition after pre-treatment. The following are the four treatment combinations: ERG ST; ERG ST+FAM; ME+ERG ST; ME+ERG ST+FAM. Four subjects will be enrolled in the study and randomized. The primary outcome is to improve emotion dysregulation in participants. Emotion dysregulation will be measured using the Difficulties in Emotion Regulation Scales (DERS).

DETAILED DESCRIPTION:
The goal of this pilot study was to carry out a randomized controlled trial to investigate whether motivational enhancement therapy (MET) improved the treatment effects of a 12-week psychological intervention, Dialectical Behaviour Therapy Skills Training (DBT-ST), for EA presenting in the early stages of mental health difficulties. Participants were recruited from the Youth Wellness Centre at St. Joseph's Healthcare Hamilton and McMaster University's Student Wellness Centre in Hamilton, Canada.

Methods: Seventy-five participants were randomized to receive MET followed by DBT-ST or to DBT-ST alone. We assessed psychological distress, emotion dysregulation, and depression and anxiety symptoms as outcomes. Results: We found that both treatment groups had significant reductions in emotional dysregulation, psychological distress, depression, and anxiety at post- treatment and at the 3-month follow-up. Participants assigned to MET pre-treatment experienced greater improvement in psychological distress at the end of treatment. Conclusion: This pilot study provides preliminary evidence of the potential augmentation of DBT-ST using MET in a real-world setting. Future studies should examine whether MET uniquely augments DBT-ST through the use of a comparable pre-treatment control group.

ELIGIBILITY:
Inclusion Criteria:

1. Help-seeking youth (ages 17-25 years)
2. Literacy in English
3. Early stage mental health concerns of mild to moderate severity
4. Emotional dysregulation

Exclusion Criteria:

1. Diagnosis of Borderline Personality Disorder
2. Diagnosis of Anorexia Nervosa or Bulimia Nervosa
3. Diagnosis of Posttraumatic Stress Disorder (current)
4. Moderate to Severe Depression (current)
5. Bipolar Disorder and related disorders
6. Diagnosis of Schizophrenia and other psychotic disorders
7. Diagnosis of Antisocial Personality Disorder (ASPD)
8. DSM-5 Substance Use disorder of Moderate or Severe severity (current)
9. Moderate to Severe Self-Harm behaviour within past year
10. Hospital admission for mental health concerns within past 6 months
11. Multiple (2+) Psychiatric Emergency Service visits within past 6 months

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Emotion Regulation throughout 12-week ERG group, at post ERG group and 16-week follow-up to group. | Baseline (2 weeks pre-ERG ST), Weeks 1, 4, 9 and 12 of ERG ST and 12 weeks after the end of ERG ST
  The Difficulties in Emotion Regulation Scales is a 36-item self-report measure of emotion dysregulation with adequate psychometric properties.

SECONDARY OUTCOMES:
GAIN-Q3-MI-ONT | Baseline (2 weeks pre-ERG ST) and post-treatment (week 12 of ERG-ST)
  The GAIN-Q3-MI-ONT includes the following scales: School Problems, Work Problems, Health Problems, Sources of Stress, Risk Behaviours, Internalizing Disorders, Externalizing Disorders, Substance Disorders, Crime & Violence and Total Disorder. For most individual screeners, internal consistency is good to excellent (alpha > .7) for adolescents and adults.
Sheehan Disability Scale | Baseline (2 weeks pre-ERG ST), Weeks 1, 4, 9 and 12 of ERG ST and 12 weeks after the end of ERG ST
  Functioning will be measured using the Sheehan Disability Scale, a self-report measure of functioning in: home, work/school, and the social realm.
Kessler Psychological Distress Scale (K-10) | Baseline (2 weeks pre-ERG ST), Weeks 1, 4, 9 and 12 of ERG ST and 12 weeks after the end of ERG ST
  Psychological distress will be measured using the K-10, a brief and well-validated instrument.
Dialectical Behaviour Therapy Ways of Coping Checklist (DBT-WCCL) | Baseline (2 weeks pre-ERG ST), Weeks 1, 4, 9 and 12 of ERG ST and 12 weeks after the end of ERG ST
  The DBT-WCCL which has adequate validity and reliability, will be used as a measure of coping skills.
The Depression Anxiety and Stress Scales 21 (DASS-21) | Baseline (2 weeks pre-ERG ST), Week 12 of ERG ST and 12 weeks after the end of ERG ST
  The Depression Anxiety and Stress Scales 21 (DASS-21) is a 21-item short-form measure of depression, anxiety and stress. Reliability, measured using Cronbach's alpha, has been shown to be adequate: alpha = .93 for the total scale. The DASS-21 has shown good convergent and discriminant validity when compared with other measures of depression and anxiety.
Burden Assessment Scale | Baseline (2 weeks pre-ERG ST), Week 12 of ERG ST and 12 weeks after the end of ERG ST
  The Burden Assessment Scale, which assesses levels of objective and subjective burden, and the Perceived Burden Scale, which assesses interpersonal burden and role strain, will be used as a measure of caregiver burden.
Modified M.I.N.I. Screener (MMS) | Baseline (2 weeks pre-ERG ST)
  The MMS is designed to identify people who need a mental health assessment, covering mood disorders, anxiety and psychotic disorders.
Lifetime Suicide Attempt Self Injury (L-SASI) | Baseline (2 weeks pre-ERG ST)
  The L-SASI is an interview to collect lifetime history details of non-suicidal self-injury and suicidal behaviour. The interview will be used to exclude individuals who have had moderate to severe self-harm within the past year.
The International Personality Disorder Examination (IPDE) | Baseline (2 weeks pre-ERG ST)
  This measure will be used to determine a probable or negative diagnosis of BPD in order to support the diagnosis of BPD exclusion criteria.
Patient Health Questionnaire (PHQ) | Baseline (2 weeks pre-ERG ST), Week 12 of ERG ST and 12 weeks after the end of ERG ST
  A diagnostic tool that will be used as a screener for depression, anxiety, eating disorders and alcohol use.
Readiness for Change | Baseline (2 weeks pre-ERG ST), Week 1 of ERG ST
  Participants will indicate their readiness to engage in treatment using the Readiness for Change questionnaire which was derived directly from the GAIN-Q3.
Validating and Invalidating Response Scale (VIRS-kids) | Baseline (2 weeks pre-ERG ST), Week 1 and 12 of ERG ST and 12 weeks after the end of ERG ST
  VIRS-kids is a measure of how much a caregiver's validation and invalidation impacts a youth's emotional regulation, behavior and care giver-youth relationship satisfaction.
The M.I.N.I. International Neuropsychiatric Interview | Baseline (2 weeks pre-ERG ST) and Week 12 of ERG ST
  This is a brief structured interview for the major psychiatric disorders in the DSM. It assesses for: major depressive episode, suicidality, manic episode, bipolar disorders, panic disorder, agoraphobia, social phobia, obsessive-compulsive disorder, posttraumatic stress disorder, alcohol abuse and dependence, substance use and dependence, psychotic disorders, anorexia nervosa, bulimia nervosa, generalized anxiety disorder. The M.I.N.I. will be used to ensure that exclusion criteria are not being met.
Borderline Symptom List 23 (BSL-23) | Baseline (2 weeks pre-ERG ST), Week 12 of ERG ST and 12 weeks after the end of ERG ST
  The BSL-23 will be used to screen for Borderline Personality Disorder (BPD) symptoms and self-harm behaviours.
Brief Treatment History Interview (B-THI) | Baseline (2 weeks pre-ERG ST), Week 12 of ERG ST and 12 weeks after the end of ERG ST
  A selection of questions from the B-THI that contains face-valid questions will be used to assess for hospitalization and psychiatric emergency use, psychotropic medication and receipt of ancillary psychotherapy.
Family Assessment Device (FAD) | Baseline (2 weeks pre-ERG ST), Week 12 of ERG ST and 12 weeks after the end of ERG ST
  FAD is a 53 item self-report measure designed to measure family function (31). The FAD is made up of seven scales which measure Problem Solving, Communication, Roles, Affective Responsiveness, Affective Involvement, Behaviour Control and General Functioning. The reliability, measured using Cronbach's alpha, ranged from 0.72 (Roles and Behaviour Control) to 0.92 (General Functioning).
Texas Grief Inventory | Baseline (2 weeks pre-ERG ST), Week 12 of ERG ST and 12 weeks after the end of ERG ST
  The Texas Grief Inventory, which has three subscales: grief (15 items), mastery (15 items) and empowerment (19 items), will be used to measure caregivers' sense of empowerment.
Adult Behaviour Checklist (ABCL) | Baseline (2 weeks pre-ERG ST), Week 12 of ERG ST and 12 weeks after the end of ERG ST
  The Adult Behaviour Checklist for ages 18-59 (ABCL) is a checklist used to obtain information on a range of mental health and substance use concerns. The family/friends will report on the youth's difficulties. Authors report internal consistency alphas ranging from 0.78 to 0.85 and test-retest reliability ranging from r = 0.73-0.92.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Zipursky, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton - Youth Wellness Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGorry PD, Purcell R, Hickie IB, Yung AR, Pantelis C, Jackson HJ. Clinical staging: a heuristic model for psychiatry and youth mental health. Med J Aust. 2007 Oct 1;187(S7):S40-2. doi: 10.5694/j.1326-5377.2007.tb01335.x. PMID 17908024
- [Background] Soler J, Pascual JC, Tiana T, Cebria A, Barrachina J, Campins MJ, Gich I, Alvarez E, Perez V. Dialectical behaviour therapy skills training compared to standard group therapy in borderline personality disorder: a 3-month randomised controlled clinical trial. Behav Res Ther. 2009 May;47(5):353-8. doi: 10.1016/j.brat.2009.01.013. Epub 2009 Jan 29. PMID 19246029